CLINICAL TRIAL: NCT04846049
Title: An Inter-Disciplinary Outpatient Care Model Providing Comprehensive Geriatric Assessment, Care-Coordination and Co-management to High Need High Risk Veterans Meeting HBPC Criteria
Brief Title: Inter-Disciplinary Outpatient Care Model Providing Comprehensive Geriatric Assessment, Care-Coordination & Co-management
Acronym: C4
Status: Completed | Type: Observational
Sponsor: Miami VA Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stuti Dang, Physician, Miami VA Healthcare System
Other Study IDs: 1208331-1
Record Dates: First submitted 2019-03-05; First posted 2021-04-15 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Veterans; Geriatric Assessment; Care-Coordination; Outpatient Care
Keywords: High Need High Risk; Home Based Primary Care
MeSH Terms: interventions — Comprehensive Health Care; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Comprehensive Care: Veterans with complex medical conditions that may need more help. This intervention will provide extra care coordination after a complete assessment of their health.
  Research team will assess veteran's memory, physical function, strength, balance, and from there, find the areas they need the most help with and coordinate services at home. This is in addition to their regular primary care provider.
  Interventions: Other: Comprehensive Care
- Standard Care: Veterans receiving standard of care
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Comprehensive Care — 1. Comprehensive Geriatric Assessment (3 visits with a geriatrician alternating with 3 primary provider visits over 6 months)
  2. Care Planning with Interdisciplinary Team
  3. Care coordination
  4. Co-management with Primary care
  5. Social work needs assessment
  6. Patient-centered telehealth using phone, home telehealth, patient portal, Video
  7. Transportation provided for all visits
  8. Referral to Geriatric primary care clinic and mental health per Veteran need
  9. Goals of Care and Veteran preferences conversation
  10. Educate primary care providers about HNHR population, home and community based services, collaboration
  Groups: Comprehensive Care
Other: Standard Care — No intervention or treatment will be provided.
  Groups: Standard Care

SUMMARY:
The Department of Veterans Affairs' (VA) Home Based Primary Care (HBPC) program provides comprehensive care to its sickest, frailest Veterans with multiple complex chronic diseases. The HBPC program is a resource intensive non-institutional care program where Veterans, who are not able to receive primary care at the VA, are closely monitored and care is provided using an interdisciplinary team that coordinates the care through multi-professional home visits.

The Geriatric Extended Care recommended that Miami Veteran Affairs Healthcare System (VAHS) HBPC enroll from a list of over 2,000 pre-identified High Need High Risk (HNHR) Miami Veterans for whom HBPC enrollment would have a high likelihood of clinical and economic benefits. HNHR Veterans have the greatest need for care but face the steepest challenges with access. However, despite best of intentions, the Miami HBPC program does not have the capacity to enroll the large numbers of Veterans on this new HNHR list. Therefore, innovative strategies are needed to provide appropriate needed care for this HNHR Veteran population.

Goal: Maintain older Veterans in their homes for as long as possible.

Aims: Design and pilot test an evidence-based, outpatient, Comprehensive geriatric assessment, Care plan based, Care-coordination, Co-management (C4) model, for 100 HBPC eligible HNHR older Veterans who are not enrolled in the HBPC program.

The investigators will develop, implement and evaluate a VA model to provide a comprehensive geriatric assessment of HNHR Veterans, design a structured care plan that includes care coordination to link their needs to appropriate referrals, home and community based services, monitor and coach patients and caregivers, and coordinate their care across VA and non-VA providers and settings.

Objectives:

1. Characterize the needs of the HNHR group of Veterans
2. Evaluate the feasibility and processes of the Geri C4 model
3. Evaluate the impact of the model on patient, healthcare utilization, and other Geriatric Extended Care (GEC) outcomes
4. Determine the facilitators and barriers for implementing the intervention

DETAILED DESCRIPTION:
The intervention will consist of the following components:

1. Comprehensive Geriatric Assessment: A complete geriatric assessment using an interdisciplinary team (geriatrician, psychologist, social worker, dietitian, and nurse). The investigators will increase the number of geriatrician and interdisciplinary team visits to every other month interspersed with their primary care visits.
2. Care Planning: The investigators will review and discuss each participant during the interdisciplinary team meeting. The team will jointly generate a care plan for the implementation of the interventions. The care plan will be shared with the respective primary care provider.
3. Care Coordination: Participant/caregiver will be regularly contacted to confirm that the care plan is being implemented and to allow the participant/caregiver to discuss issues related to the management.
4. Co-management: Primary care provider and project Geriatricians will share responsibility and decision making for participants aiming to prevent and treat geriatric complications.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in prior 12-months
* Received post-acute care in prior 12-months (skilled nursing facility or skilled home health care)
* Two or more chronic conditions
* Two or more activity of daily living impairments or greater or equal to six Frailty Index score
* Less than or equal to 60 minutes of closest VA primary care site.

Exclusion Criteria:

* Enrolled in Home Based Primary Care
* Using hospice Care
* Using palliative care
* In a foster home
* In a nursing home

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: High Need High Risk Veterans in Miami Medical Center area
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in FRAIL score | 5 minutes
  The FRAIL scale (Fatigue, Resistance, Ambulation, Illnesses, & Loss of Weight) is a simple questionnaire of frailty syndrome for older adults. If a patient scores 3-5 points over a total score of 5 points in the FRAIL, the patient is considered as frail. Change from baseline score and 6 months.
Change in Montreal Cognitive Assessment (MOCA) | 10 minutes
  Rapid screen of cognitive abilities designed to detect mild cognitive dysfunction consisting of 16 items and 11 categories assessing multiple cognitive domains. No cognitive impairment >=25 Mild cognitive impairment = 20-24 Severe cognitive impairment < 20. Change from baseline score and 6 months.

SECONDARY OUTCOMES:
Katz Index of Independence in Activities of Daily Living | 10 minutes
  Assessment of activities of daily living. Change from baseline score and 6 months.
Lawton-Brody Instrumental Activities of Daily Living Scale | 10 minutes
  Instrumental activities of daily living assessment. Change from baseline score and 6 months.
Detection of symptoms of depression | 5 minutes
  Patient Health Questionnaire (PHQ-2 and PHQ-9) for depression. The PHQ 2 is a preliminary screening tool administered before the PHQ 9. If a patient responds 'yes´ to one or both questions on the PHQ-2, the PHQ-9 questions are administered. Cut-off is set to a score of ≥ 2 PHQ-2. PHQ-9 scoring: 0-4 none-minimal; 5-9 mild;10-14 moderate; 15-19 moderately severe; 20-27 severe.
Change in number of clinic visits | 6-months
  Changes in pre intervention number of clinic visits. This will be measure by survey and chart review.
Change in number of hospital admissions | 6-months
  Changes in pre intervention number of hospital admissions. This will be measure by survey and chart review.
Change in healthcare utilization | 6-months
  Changes in pre intervention number of Home and Community Based services in place. This will be measure by survey and chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Stuti Dang, MD,MPH, Principal Investigator — Miami VA Healthcare System
Locations (1):
- Miami VA Healthcare System, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No